CLINICAL TRIAL: NCT03811171
Title: A Study of the SonoMotion Break Wave(TM) System for the Comminution of Urinary Tract Stones
Brief Title: Break Wave(TM) Extracorporeal Lithotripter First-in-Human Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SonoMotion (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-0001; R44DK109779 (NIH)
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Renal Calculi; Urinary Calculi
Keywords: Stone; Lithotripsy; Calculi
MeSH Terms: conditions — Kidney Calculi; Urinary Calculi; Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): The arm receives the investigational Break Wave procedure.
  Interventions: Device: Break Wave extracorporeal lithotripsy

INTERVENTIONS:
Device: Break Wave extracorporeal lithotripsy — The Break Wave device will be used to exert a low amplitude burst of ultrasound waves focused at the kidney stone. The primary components of the device include an 85 mm aperture diameter therapy probe driven by a high voltage generator. The therapy probe has a cavity in the middle to accommodate coaxial alignment of an ultrasound imaging probe for treatment guidance.

SUMMARY:
This is a prospective, open-label, multi-center, single-arm (non-randomized) study to assess the safety and effectiveness of breaking stones in the upper urinary tract using the SonoMotion Break Wave technology. Up to 30 subjects will be included. The procedure will be performed in a hospital surgical environment as an outpatient (without being admitted) or in a non-surgical environment such as a clinic or office procedure room. The procedure will be performed under varying levels of anesthesia ranging from no anesthesia to general anesthesia (fully asleep). Stones will be limited to ≤ 10 mm for lower pole stones and ≤ 20 mm everywhere else.

Safety will be measured by the self-reported occurrences of adverse events, unplanned emergency department or clinic visits, and the need for further intervention. Fragmentation will be measured by self-reported stone passage and a comparison of computed tomography (CT) images before and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Individuals presenting with at least one kidney stone apparent on CT.
* Stones must be within the upper urinary tract.
* Stones are indicated for SWL treatment per the American Urology Association (AUA) 2016 guidelines.8
* Stones must be measured under CT to be within the AUA 2016 SWL guidelines (i.e. ≤ 10 mm for lower pole stones and ≤ 20 mm for non-lower pole stones).

Exclusion Criteria:

* Acute untreated urinary tract infection or urosepsis.
* Uncorrected bleeding disorders or coagulopathies.
* Pregnancy.
* Uncorrected obstruction distal to the stone.
* Patients receiving anticoagulants and who are unable or not willing to cease the medication for the Break Wave procedure.
* Stones that are not echogenically visible or cannot be positioned within the Break Wave therapy focus.
* Individuals belonging to a vulnerable group (pregnant, mentally disabled, prisoner, etc.).
* Patients unwilling to comply with the follow-up protocol, including post-procedure CT.
* Individuals under 18 years of age.
* Anatomic presentations preventing adequate positioning or delivery of the Break Wave pulse.
* Calcified abdominal aortic aneurysms or calcified renal artery aneurysms.
* Solitary kidney
* Comorbidity risks which, in at the discretion of the physician, would make the patient a poor candidate for the Break Wave procedure, such as anatomical anomalies that may not be conducive to adequate stone fragment passage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Outcome - Stone Fragmentation | 12 weeks post-treatment
  Stone fragmentation as determined by stone passage or imaging confirmation.
Primary Safety Outcome - Hematoma, urinary tract sepsis, or cardiac arrythmia | 12 weeks post-treatment
  The documented occurrence of clinically significant or symptomatic hematoma (perirenal/intrarenal), urinary tract sepsis, or serious cardiac arrythmia.

SECONDARY OUTCOMES:
Secondary effectiveness outcome - Stone Free Status | 12 weeks post-treatment
  Radiographic evidence (CT imaging) of stone free status.
Secondary effectiveness outcome - Residual fragment size | 12 weeks post-treatment
  Presence of only stone fragments small enough to pass (less than or equal to 4 mm).
Secondary safety outcome - Adverse events | 12 weeks post-treatment
  documented occurrence of all adverse events and comparison of the incidence (rate of occurrence) to the adverse events associated with shock wave lithotripsy (SWL)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - University of California San Diego Health, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of Washington Medical Center, Seattle, Washington
- Canada (3):
  - University of Alberta, Division of Urology, Edmonton, Alberta
  - Vancouver General Hospital Stone Centre, Vancouver, British Columbia
  - St. Michael's Unity Health Toronto, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chew BH, Harper JD, Sur RL, Chi T, De S, Buckley AR, Paterson RF, Wong VKF, Forbes CM, Hall MK, Kessler R, Bechis SK, Woo JR, Wang RC, Bayne DB, Bochinski D, Schuler TD, Wollin TA, Samji R, Sorensen MD. Break Wave Lithotripsy for Urolithiasis: Results of the First-in-Human International Multi-Institutional Clinical Trial. J Urol. 2024 Oct;212(4):580-589. doi: 10.1097/JU.0000000000004091. Epub 2024 Sep 10. PMID 39254129
- [Background] Maxwell AD, Cunitz BW, Kreider W, Sapozhnikov OA, Hsi RS, Harper JD, Bailey MR, Sorensen MD. Fragmentation of urinary calculi in vitro by burst wave lithotripsy. J Urol. 2015 Jan;193(1):338-44. doi: 10.1016/j.juro.2014.08.009. Epub 2014 Aug 9. PMID 25111910
- [Background] Maxwell AD, MacConaghy B, Bailey MR, Sapozhnikov OA. An investigation of elastic waves producing stone fracture in burst wave lithotripsy. J Acoust Soc Am. 2020 Mar;147(3):1607. doi: 10.1121/10.0000847. PMID 32237849
- [Background] Sapozhnikov OA, Maxwell AD, Bailey MR. Modeling of photoelastic imaging of mechanical stresses in transparent solids mimicking kidney stones. J Acoust Soc Am. 2020 Jun;147(6):3819. doi: 10.1121/10.0001386. PMID 32611160
- [Background] Harper JD, Lingeman JE, Sweet RM, Metzler IS, Sunaryo PL, Williams JC Jr, Maxwell AD, Thiel J, Cunitz BW, Dunmire B, Bailey MR, Sorensen MD. Fragmentation of Stones by Burst Wave Lithotripsy in the First 19 Humans. J Urol. 2022 May;207(5):1067-1076. doi: 10.1097/JU.0000000000002446. Epub 2022 Mar 21. PMID 35311351
- See also: Sponsor Website — http://www.sonomotion.com